CLINICAL TRIAL: NCT01290614
Title: A Chronic Care Model Based QI Program to Improve the Care of Patients With CKD
Brief Title: A Chronic Care Model Based Quality Improvement (QI) Program to Improve the Care of Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10088-H41
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist intervention (Experimental)
  Interventions: Other: Pharmacist based QI program
- Control - usual care (Active Comparator): Patients assigned to control will continue to receive care from their VA provider.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Pharmacist based QI program — Per a study protocol, the pharmacist will call each subject (who has not opted out) and discuss their CKD. In brief, the pharmacist will introduce themselves, ask the subject if they have time to discuss their medical care, inform the subject that they have CKD, briefly discuss CKD, ask the subject if they can come for labs, discuss hypertension management as appropriate, and answer any questions. In addition, for subjects with poorly controlled hypertension, the study pharmacist will arrange for a nutrition consult for a low sodium diet, a mainstay of hypertension management in patients with CKD. Finally, for patients with advanced CKD (GFR <30 mL/min per 1.73 m2) who are not seeing a nephrologist, the study pharmacist will arrange for a nephrology outpatient appointment to assess the need for placement of access for renal replacement therapy.
  Arms: Pharmacist intervention
Other: Usual Care — Patients in the control arm will continue to receive "usual care" from their VA providers.
  Arms: Control - usual care

SUMMARY:
The goal of this study is to evaluate the impact of a chronic care model (CCM) based quality improvement program on 1) outcomes for patients with chronic kidney disease (CKD) and 2) adherence to CKD guidelines. This pilot study will evaluate the feasibility of a CCM based quality improvement program for patients with CKD and assess potential mechanisms for the intervention's effect.

Hypothesis: Implementing a CCM based quality improvement program including system level support in the form of collaborative care, a CKD registry, and provider education will 1) reduce systolic BP in patients with poorly controlled hypertension, 2) increase the percentage of patients appropriately monitored for metabolic complications, and 3) decrease the rate of catheter use in patients initiating dialysis.

DETAILED DESCRIPTION:
Research Plan:

The experimental design is a prospective, randomized controlled trial evaluating the impact of a Chronic Care Model (CCM) based quality improvement program on CKD guideline adherence. The intervention will focus on three main goals: 1) reduction of BP to target levels, 2) appropriate monitoring of patients for metabolic complications of CKD, and 3) reduced use of dialysis catheters in patients initiating dialysis. The CKD CCM QI program will include a lecture on CKD guidelines and hypertension to all CBOC providers and a centrally located pharmacist with access to the CKD registry.

Methodology:

Veterans receive primary care at Community Based Outpatient Centers (CBOCs) throughout Northeast Ohio. Patients with CKD who receive their primary care at a Northeast Ohio CBOC will be eligible for the study. The hypothesis was formulated before data collection.

ELIGIBILITY:
Inclusion Criteria:

* receipt of primary care at a VISN 10 Northeast Ohio CBOC
* GFR (calculated according to the 4 variable Modification of Diet in Renal Disease study equation) less than 45 mL/min per 1.73m2 with a second GFR less than 60 at least 90 to 730 days prior to the index GFR (26); and
* at least one primary care visit in the year prior to study initiation.

Exclusion Criteria:

* ESRD as defined by chronic renal replacement therapy,
* receipt of a renal transplant,
* hospice care, and
* age greater than 85 years or less than 18 years at the time of study initiation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2199 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Drawz, MD, MHS, MS, Principal Investigator — LSCDVAMC
Locations (1):
- LSCDVAMC, Cleveland, Ohio, United States

REFERENCES:
- [Result] Cooney D, Moon H, Liu Y, Miller RT, Perzynski A, Watts B, Drawz PE. A pharmacist based intervention to improve the care of patients with CKD: a pragmatic, randomized, controlled trial. BMC Nephrol. 2015 Apr 16;16:56. doi: 10.1186/s12882-015-0052-2. PMID 25881226
- [Derived] Campbell ZC, Dawson JK, Kirkendall SM, McCaffery KJ, Jansen J, Campbell KL, Lee VW, Webster AC. Interventions for improving health literacy in people with chronic kidney disease. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD012026. doi: 10.1002/14651858.CD012026.pub2. PMID 36472416
- See also: Open Access version of manuscript — http://www.biomedcentral.com/1471-2369/16/56

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacist Intervention | Control - Usual Care
Started | 1070 | 1129
Completed | 518 | 1129
Not Completed | 552 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist Intervention | Control - Usual Care | Total
Number analyzed (Participants) | 1070 | 1129 | 2199
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (8.2) | 75.7 (8.2) | 75.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 1054 | 1106 | 2160
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 62 | 56 | 118
  Not Black | 1008 | 1073 | 2081
Region of Enrollment [Number; unit: participants]
  United States | 1070 | 1129 | 2199

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure (SBP)
Description: Average SBP for those with a baseline BP > 130/80
Time Frame: one year
Population: Baseline blood pressure >130/80 mmHg
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pharmacist Intervention | Control - Usual Care
Number analyzed (Participants) | 474 | 473
mmHg | 135.1 (17.4) | 134.4 (17.6)
Statistical Analysis 1: Comparison: Pharmacist Intervention vs Control - Usual Care; Test type: Superiority or Other; p = 0.57, t-test, 2 sided

2. Secondary Outcome: Number of Participants With PTH Measurement During the Study Period
Description: The primary process outcome was measurement of PTH during the study period.
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Pharmacist Intervention | Control - Usual Care
Number analyzed (Participants) | 1070 | 1129
participants | 502 | 182
Statistical Analysis 1: Comparison: Pharmacist Intervention vs Control - Usual Care; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Pharmacist Intervention | Control - Usual Care
Serious Adverse Events (participants affected / at risk) | 0/1070 | 0/1129
Other Adverse Events (participants affected / at risk) | 0/1070 | 0/1129

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No